CLINICAL TRIAL: NCT02560532
Title: A Prospective, Multi-center, Open-label, Single-arm, Phase 2 Study to Assess the Efficacy and Safety of Clazosentan in Reversing Angiographically-confirmed Cerebral Vasospasm in Adult Subjects With Aneurysmal Subarachnoid Hemorrhage (aSAH) Treated by Surgical Clipping or Endovascular Coiling
Brief Title: Evaluation of the Efficacy and Safety of Clazosentan in Reversing Cerebral Vasospasm in Adult Subjects With Aneurysmal Subarachnoid Hemorrhage
Acronym: REVERSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-054-203; 2015-002721-18 (EudraCT Number)
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysmal subarachnoid hemorrhage; cerebral vasospasm; clazosentan
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — clazosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clazosentan (Experimental): Diluted solution administered as a continuous intravenous infusion at a rate of 15 mg/h for up to a cumulative maximum of 10 days
  Interventions: Drug: Clazosentan

INTERVENTIONS:
Drug: Clazosentan — Concentrated solution for intravenous injection
  Other Names: ACT-108475

SUMMARY:
The purpose of this study is to evaluate the safety and potential therapeutic benefit of use of clazosentan in reversing cerebral vasospasm (a narrowing of blood vessels in the brain due to the presence of blood in the space around the brain) in patients who have suffered a condition known as aneurysmal subarachnoid hemorrhage caused by bleeding onto the surface of the brain from a ruptured brain aneurysm

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is characterized by bleeding onto the brain surface due to a rupture of a pouch or bulge in a brain vessel (called an aneurysm). It is a rare but serious condition with a high risk of death. Even patients who have had successful repair of the aneurysm remain at risk for developing cerebral vasospasm, which can result in harmful conditions related to the lack of oxygen to parts of the brain and death. Cerebral vasospasm usually occurs within the first couple of weeks after aSAH, and it is difficult to treat. Currently there is no safe, efficacious and widely available treatment. Previous animal studies have shown that a new drug under investigation, clazosentan, was able to reverse cerebral vasospasm in animal models of SAH. A first trial conducted in a small number of patients showed some benefit of clazosentan in reversing established cerebral vasospasm after aSAH. Clazosentan has already been evaluated in the prevention of cerebral vasospasm in several large clinical trials in aSAH. This current study aims to evaluate if clazosentan is effective and safe in the treatment of cerebral vasospasm after aSAH.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from the subject or proxy/legal representative
* Aneurysmal subarachnoid hemorrhage (aSAH)confirmed by digital subtraction angiogram (DSA) or computed tomography angiogram (CTA), successfully secured by surgical clipping or endovascular coiling within 72 hours of rupture
* World Federation of Neurological Surgeons (WFNS) grade 1-4 at admission, and which must not increase to grade 5 at the time of enrollment
* Moderate or severe global cerebral vasospasm at the time of enrollment, documented by digital subtraction angiography (DSA) performed not earlier than 48 hours post aneurysm-securing procedure
* Women of childbearing potential must have a negative serum pregnancy test at screening and must use a reliable method of contraception from hospital discharge up to 30 days after discontinuation of study drug infusion, and fertile males must use a condom as a contraceptive method during this same period

Exclusion Criteria:

* SAH due to causes other than a saccular aneurysm
* Any moderate or severe cerebral vasospasm on angiography prior to the aneurysm-securing procedure
* Presence of a new or worsened cerebral infarct or evidence of significant bleeding post aneurysm-securing procedure, or re-bleeding, on a CT scan performed within 24 hours prior to enrollment
* Total bilirubin > 2 times the upper limit of normal, and / or a known diagnosis or clinical suspicion of liver cirrhosis or moderate to severe hepatic impairment
* Any severe or unstable concomitant condition or disease (e.g., cancer, hematological, or coronary disease) or chronic condition (e.g., drug abuse, severe alcoholism), which, in the opinion of the investigator, would interfere with the assessment of the safety or effect of the study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-01; Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Successful reversal of global cerebral vasospasm 3 hours post-study drug initiation | 3 hours post-study drug initiation
  Successful reversal is defined as an improvement in at least one level of severity on the "global vasospasm assessment" (i.e., from severe to moderate, mild, or none, or from moderate to mild or none), evaluated on Digital subtraction angiogram (DSA)

SECONDARY OUTCOMES:
Successful reversal of global cerebral vasospasm 24 hours post-study drug initiation | 24 hours post-study drug initiation
Maximum change from baseline in angiographic cerebral circulation time (CCT) | At baseline, 3 hours and 24 hours post-study drug initiation
  CCT will be determined in the left and right anterior circulation, and the posterior circulation, on the digital subtraction angiogram (DSA) at each scheduled time point.
Number of subjects with adverse events | Up to 30 days after study drug discontinuation
  An adverse event is defined as any unfavorable and unintended sign, including an abnormal laboratory finding, symptom or disease, that occurs during the course of the study, whether or not considered related to the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Marr, BSc. Pharm, Study Director — Actelion
Locations (11):
- Site 2002, Helsinki, Finland
- France (5):
  - Site 1002, Bron
  - Site 1006, Clermont-Ferrand
  - Site 1004, Marseille
  - Site 1005, Montpellier
  - Site 1001, Paris
- Switzerland (5):
  - Site 3005, Aarau
  - Site 3001, Basel
  - Site 3003, Bern
  - Site 3004, Geneva
  - Site 3002, Zurich